CLINICAL TRIAL: NCT06931171
Title: Zero-cost Radiation Protection Method to Reduce Radiation Exposure of Interventional Cardiologists During Transradial Percutaneous Coronary Procedures (FREEPADRAD Trial)
Acronym: FREEPADRAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Georgios Latsios, Director of Cardiology, Principal Investigator, Interventional Cardiologist, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FREEPADRAD
Record Dates: First submitted 2025-02-13; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Occupational Radiation Exposure in Interventional Cardiology
Keywords: Occupational Radiation Exposure; Interventional Cardiology; Radiation Protection; Transradial Access; Radiation Safety; Operator Radiation Dose; Radiation Hazard Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Use of conventional radiation protection measures. (No Intervention): This group will undergo transradial coronary procedures using only conventional radiation protection measures. These include standard operator lead aprons, fixed protective drapes, and other standard shielding equipment typically employed in the catheterization laboratory. No additional radiation protection devices or techniques will be applied to the patient. This arm serves as the baseline for comparison with the intervention group.
- Additional patient-applied pelvic lead shielding (Experimental): This group will undergo transradial coronary procedures with the addition of a patient-applied pelvic lead shield. Alongside the conventional radiation protection measures used in the control group, a triple-layer lead apron will be placed over the patient's lower abdominal and pelvic region. This shield, composed of three 0.25 mm Pb-equivalent layers, is designed to reduce scatter radiation exposure to the operator. The intervention aims to assess the effectiveness of this additional protective measure in reducing operator radiation dose.
  Interventions: Radiation: Patient-Applied Pelvic Lead Shielding

INTERVENTIONS:
Radiation: Patient-Applied Pelvic Lead Shielding — The intervention involves the application of a triple-layer lead apron to the patient's lower abdominal and pelvic region during transradial coronary procedures. The apron measures 75 cm × 45 cm and is composed of three layers of 0.25 mm Pb-equivalent material. This protective shield is placed on the patient in addition to standard operator radiation protection measures. The primary goal of this intervention is to reduce scatter radiation exposure to the operator, thereby improving occupational safety in the catheterization laboratory. This approach leverages existing radiation protection materials in a novel configuration.
  Arms: Additional patient-applied pelvic lead shielding

SUMMARY:
Ionising radiation is a recognised occupational hazard in interventional cardiology. This prospective, randomised trial aims to evaluate the effectiveness of additional radiation protection by existing devices but with a different use, specifically the use of medical lead aprons (designed and used to be worn by the medical and nursing staff for radiation protection) covering the patient's lower abdominal and pelvic area during transradial coronary angiography and angioplasty. The intervention's efficacy will be assessed by measuring the reduction in operator radiation exposure and determining the impact of various clinical and procedural factors.

DETAILED DESCRIPTION:
Ionizing radiation refers to any type of radiation capable of interacting with matter. It plays a vital role in medical diagnostics and therapeutic applications. Imaging techniques allow for timely and accurate diagnosis, while advanced therapies contribute to longer life expectancy and improved quality of life. However, ionizing radiation carries inherent risks, making its controlled use essential. Radiation exposure is not immediately perceptible but can result in significant damage to the exposed organism. Common effects of high-dose exposure include ocular damage and skin injuries, while radiation is also associated with cellular-level damage, leading to an increased risk of malignancies. Exposure is proportional to time, inversely proportional to the square of the distance from the source, and accumulates over time.

Despite technological advancements and improved X-ray systems, the increasing complexity and frequency of interventional cardiology procedures have led to higher radiation exposure in catheterization laboratories. This poses a major occupational hazard for medical staff, highlighting the need for effective methods to reduce radiation exposure and protect healthcare professionals. Operator radiation exposure varies depending on experience, procedure type, patient characteristics, X-ray system features, and protective measures used. These measures include disposable gloves, shields, lead aprons, and robotic systems.

This prospective, randomised trial evaluates the efficacy of a cost-effective (namely zero-cost) and very easily utilised radiation protection strategy for interventional cardiologists during transradial coronary procedures. By applying a triple-layer lead apron to the patient's pelvic region, the study aims to reduce operator radiation exposure while maintaining standard procedural outcomes. The randomized controlled trial will compare the intervention group utilizing the additional shielding with a control group employing standard radiation protection methods. Key measurements include direct operator radiation exposure and its relation to patient-specific and procedural factors. Findings may establish a practical method for reducing the specific radiation-related occupational hazard related to modern transracial interventional cardiology.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing transradial diagnostic coronary angiography or angioplasty.
* Adults aged 18 years and older.
* Informed consent provided.

Exclusion Criteria:

* Acute STEMI requiring primary percutaneous coronary intervention (PCI).
* Patients undergoing structural heart interventions.
* Initially femoral access or crossover to femoral access procedures.
* Patients unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Patient-Applied Pelvic Shielding in Reducing Operator Radiation Exposure During Transradial Coronary Procedures | During the transradial coronary procedure, measured from the start to the completion of fluoroscopy.
  Primary Outcomes:
  Absolute Operator Radiation Exposure:
  Direct measurement of operator exposure (µSv) using a dosimeter placed outside the lead apron at chest level.
Effectiveness of Patient-Applied Pelvic Shielding in Reducing Operator Radiation Exposure During Transradial Coronary Procedures | During the transradial coronary procedure, measured from the start to the completion of fluoroscopy.
  Primary Outcomes:
  Relative Operator Radiation Exposure:
  Measured as the ratio of operator exposure (µSv) to patient radiation dose area product (cGy·cm²).

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - First Department of Cardiology, Hippokration General Hospital of Athens, Athens, Attica
  - First Department of Cardiology, National and Kapodistrian University of Athens, Hippokration General Hospital of Athens, Athens, Attica

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah RM, Patel D, Abbate A, Cowley MJ, Jovin IS. Comparison of transradial coronary procedures via right radial versus left radial artery approach: A meta-analysis. Catheter Cardiovasc Interv. 2016 Dec;88(7):1027-1033. doi: 10.1002/ccd.26519. Epub 2016 Apr 1. PMID 27037544
- [Background] Vijayalakshmi K, Kelly D, Chapple CL, Williams D, Wright R, Stewart MJ, Hall JA, Sutton A, Davies A, Haywood J, de Belder MA. Cardiac catheterisation: radiation doses and lifetime risk of malignancy. Heart. 2007 Mar;93(3):370-1. doi: 10.1136/hrt.2006.098731. No abstract available. PMID 17322516
- [Background] Gutierrez-Barrios A, Camacho-Galan H, Medina-Camacho F, Canadas-Pruano D, Jimenez-Moreno A, Calle-Perez G, Vazquez-Garcia R. Effective Reduction of Radiation Exposure during Cardiac Catheterization. Tex Heart Inst J. 2019 Jun 1;46(3):167-171. doi: 10.14503/THIJ-17-6548. eCollection 2019 Jun. PMID 31708696
- [Background] Sciahbasi A, Piccaluga E, Sarandrea A, Nucci G, Caretto N, Rigattieri S, Fedele S, Romano S, Penco M. Operator Pelvic Radiation Exposure During Percutaneous Coronary Procedures. J Invasive Cardiol. 2018 Feb;30(2):71-74. Epub 2017 Dec 15. PMID 29245152
- [Background] Anadol R, Brandt M, Merz N, Knorr M, Ahoopai M, Geyer M, Krompiec D, Wenzel P, Munzel T, Gori T. Effectiveness of additional X-ray protection devices in reducing scattered radiation in radial intervention: the ESPRESSO randomised trial. EuroIntervention. 2020 Oct 23;16(8):663-671. doi: 10.4244/EIJ-D-19-00945. PMID 32338611
- [Background] Venneri L, Rossi F, Botto N, Andreassi MG, Salcone N, Emad A, Lazzeri M, Gori C, Vano E, Picano E. Cancer risk from professional exposure in staff working in cardiac catheterization laboratory: insights from the National Research Council's Biological Effects of Ionizing Radiation VII Report. Am Heart J. 2009 Jan;157(1):118-24. doi: 10.1016/j.ahj.2008.08.009. PMID 19081407